CLINICAL TRIAL: NCT02554565
Title: Innovation for Standard Identification for Insertional HPV Mutations and of Target Therapeutic Genes in Cervical Cance: Towards Development of Personalized Biomarkers in Clinical Oncology (PAIR HPV : Human PapillomaVirus)
Brief Title: Innovation for Standard Identification of Insertional HPV Mutations and of Target Therapeutic Genes in Cervical Cancer: Towards Development of Personalized Biomarkers in Clinical Oncology (PAIR HPV)
Acronym: PAIR HPV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study in competition with another so it was decided to stop recruitment
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2013-06
Record Dates: First submitted 2015-07-01; First posted 2015-09-18 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2019-03

CONDITIONS: Cervical Cancer
Keywords: Patients with cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor biopsies and blood sampling (Other)
  Interventions: Procedure: Tumor biopsy; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Tumor biopsy — Tumor biopsy before treatment
Procedure: Blood sampling — Blood sample before, during and after treatment

SUMMARY:
Quantification and follow-up of circulating tumoral DNA in serum and/or plasma of patients with cervical cancer compared to the early detection of minimal metastatic disease.

DETAILED DESCRIPTION:
Quantification and follow-up of circulating tumoral DNA in serum and/or plasma of patients with cervical cancer compared to the early detection of minimal metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with cervical cancer, at any stage, before any anti-tumoral treatment.
2. Age ≥ 18 years.
3. Patient information and signature of the informed consent or her/his legal representative.
4. Patient having given her/his agreement for a second biopsy at diagnosis if the first one was performed outside of the center and was not cryopreserved.

Exclusion Criteria:

1. Person deprived of liberty or under supervision.
2. Inability to attend scheduled follow-up visits for any psychological, sociological or geographical reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Quantification and follow-up of circulating tumoral DNA in serum and/or plasma of patients with cervical cancer compared to the early detection of minimal metastatic disease. | Until 2 years after treatment
  Detection rate of circulating tumoral DNA with confidence interval of 95% of this rate.
  Description of the variability of this rate according to the initial stage of the disease, treatment and disease progression.

SECONDARY OUTCOMES:
Validation of NGS methodology for the molecular characterization of genetic alterations related to the integration of viral DNA sequences. | Until 2 years after treatment
  Correlation between the two PCR/NGS detection methods - appreciation of the NGS method sensitivity compared to the PCR.
Detailed molecular characterization of genes alterations implicated in cervical oncogenesis. | Until 2 years after treatment
  The characterization of HPV types and HPV integration sites as well as the sequencing of representative panel of genes involved in the tumorigenesis pattway.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Besançon, Besançon
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: No